CLINICAL TRIAL: NCT01297361
Title: The Association Between Religious Origin and Age, and Vitamin B12 and Folic Acid Plasma Levels in Non Jewish Population in Western Galilee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K.Hassan
Record Dates: First submitted 2011-01-02; First posted 2011-02-16 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Vitamin B12 Deficiency; Folic Acid Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency; Folic Acid Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plasma Vitamin B12 and Folic acid levels (Other): Blood sample was drawn
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — Blood sampling for diagnosis of vitamins deficiencies

SUMMARY:
Vitamin B12 deficiency is more widespread in the population than has been assumed so far. Since a deficiency in this vitamin can lead to irreversible neurological damage, early diagnosis is essential. Vitamin B12 is synthesized exclusively in micro-organisms, and in humans it is an essential component in methyl group transfer and cell division. The vitamin is crucially involved in the proliferation, maturation, and regeneration of neural cells. In combination with folic acid, as an enzymatic essential cofactor in the metabolism of homocysteine, vitamin B12 maintains low homocysteine levels. The aim of the present study is to investigate the relationship between religious origin and age, and Vitamin B12 and Folic acid plasma levels in non Jewish population in Western Galilee. The investigators assumption is that the results of the study will contribute to early detection and treatment of Vitamin B12 and Folic acid deficiencies in order to prevent long term complications.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 and older
* Able to understand and to sign informed consent

Exclusion Criteria:

* Gastrointistinal Diseases
* Malignancy
* Psychiatric disorders
* Pregnancy
* Treatment with Vit B12 or Folic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The number of participants of each religious origin group with folic acid deficiency | 10 months
  The association between religious origin (Christians,Muslims and Druze) and folic acid plasma levels will be investigated by one blood analysis taken once at commence of trial (Day 1). Patients found to have low levels of this vitamin will be treated accordingly.
The number of participants of each age group with Vitamin B12 deficiency | 10 months
  The association between age groups (18-40, 41-65 and above 65 years old) and Vitamin B12 plasma levels will be investigated by one blood analysis taken once at commence of trial (Day 1). Patients found to have low levels of this vitamin will be treated accordingly
The number of participants of each age group with folic acid deficiency | 10 months
  The association between age groups (18-40, 41-65 and above 65 years old) and folic acid plasma levels will be investigated by one blood analysis taken once at commence of trial (Day 1). Patients found to have low levels of this vitamin will be treated accordingly
The number of participants of each religious origin group with Vitamin B12 deficiency | 10 months
  The association between religious origin (Cristians, Muslims and Druze) and Vitamin B12 plasma levels will be investigated by one blood analysis taken once at commence of trial (Day 1). Patients found to have low levels of these vitamins will be treated accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit health services, Kfar Yassif, Israel